CLINICAL TRIAL: NCT00932386
Title: The Effects of Dexmedetomidine on Tourniquet Pain Associated With Lower Extremity Surgeries Under General Anesthesia in Same Day Elective Patients
Brief Title: Effects of Dexmedetomidine on Tourniquet Pain Associated With Lower Extremity Surgeries Under General Anesthesia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: unable to secure funding for analysis of laboratory data.
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0120090056
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Orthopedic/Podiatry Procedures
Keywords: Lower extremity surgery with tourniquet use
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine Hcl infusion (Experimental): Dexmedetomidine is a highly selective alpha-2 adrenoreceptor agonist, which possesses hypnotic, sedative, anxiolytic, sympatholytic and analgesic properties.
  Interventions: Drug: Dexmedetomidine Hcl infusion
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine Hcl infusion — 0.5mcg/kg/hr
  Other Names: Precedex
  Arms: dexmedetomidine Hcl infusion
Drug: normal saline — 0.9% normal saline infusing
  Arms: normal saline

SUMMARY:
This study is being done to determine if the drug known as dexmedetomidine improves the way we care for patients when their surgery involves the use of a tourniquet on the leg. A tourniquet is sometimes used for lower leg or foot surgery to decrease the blood loss for the patient and to make it easier for the surgeon to do his work.

DETAILED DESCRIPTION:
The study will be a prospective, randomized, double blinded, and placebo controlled clinical trial. The subject population will consist of patients ages 18 to 80 undergoing same day, lower extremity surgery involving the use of a tourniquet with a minimal surgical time of 60 minutes. Subjects will be recruited on the day of surgery, after consultation with the primary surgeon as to the use of a tourniquet and the anticipated tourniquet time. Subjects will be approached while awaiting surgery either on E yellow or Same day Surgery in the Doctor's Office Complex. The study will be explained. The subject and family members will be given an opportunity to ask questions and if agreeable the subject will be asked to provide written consent. Standard American Society of Anesthesiologists monitors will be used including pulse oximetry, electrocardiogram, and non-invasive blood pressure monitoring. Both groups will have an infusion running.

The experimental group (n= 40) will have a Dexmedetomidine infusion at 0.5 mcg/kg/hr without a loading dose. The control group (n= 40) will have an equivalent volume of 0.9% normal saline infusing.

Induction will commence after the initiation of the infusion and will be identical for both groups: Midazolam 2mg IV, Fentanyl 1-2 micrograms/kg, Lidocaine 1mg/kg, and Propofol 1.5 to 2 mg/kg. Following induction an appropriately sized Laryngeal Mask Airway (LMA) will be placed. A second intravenous line (preferably 18Gauge or larger) will be placed in the opposite upper extremity to collect blood samples. Prior to sampling a waste of 10milliLiters will be withdrawn and later returned to the patient. Anesthesia will be maintained with isoflurane at a Minimum Alveolar Concentration of 0.8 to 1.2. Mean arterial pressures that exceeds 130mmHg or >30% above baseline or heart rate(HR)s >110 bpm will first be treated with additional doses of Fentanyl every two minutes for a total dose of 5mcg/kg. If there is no response following the total dose of Fentanyl then within two minutes further treatment with Labetalol consisting of titrated doses starting at 5mg IV. Rescue doses of Hydralazine up to 20mg are allowed to treat hypertension not responsive to Fentanyl and Labetalol

Measurements:

The following measurements will be collected. Time 0 : In Operating Room holding area Baseline MAP, Heart Rate(HR) , and Respiratory Rate (RR) will be recorded A baseline Numeric Ration Scale Pain Score determined

Time 1: Following Induction and prior and to tourniquet inflation MAP, HR, and RR will be recorded at five minute intervals throughout the surgical procedure

Blood samples will be analyzed for markers of stress response at four intervals.

Time 1 Following induction and prior to tourniquet inflation

Blood samples will be collected:

* C reactive Protein
* Insulin
* Cortisol
* Glucose Time 2 60 minutes after tourniquet inflation

Blood samples will be collected:

* C reactive Protein
* Insulin
* Cortisol
* Glucose

Time 3 120 minutes after tourniquet inflation or prior to tourniquet release (whichever occurs first)

Blood samples will be collected:

* C reactive Protein
* Insulin
* Cortisol
* Glucose

Time 4 30 minutes after tourniquet release

Blood samples will be collected:

* C reactive Protein
* Insulin
* Cortisol
* Glucose

Blood (15ml) will be collected from an intravenous line placed after induction of anesthesia at four time points: (1) (pre-tourniquet placement), (2) 60 minutes following inflation of the tourniquet and (3 ) 120 minutes after tourniquet inflation, and (4)approximately 30 minutes following tourniquet removal. These specimens will be placed into Vacutainer tubes with no anti-coagulant. They will be labeled with study name, subject's study ID number, sample number (1, 2, 3, 4), and date. Bloods from the first three time points will be kept refrigerated until the final sample is obtained Intra-operatively additional doses of Fentanyl and doses of Labetalol and Hydralazine will be recorded. The use of a nerve block will be documented as well.

In the Post Anesthesia Care Unit (PACU), additional doses of pain medication, anti-hypertensive medications and medications administered for relief of post operative nausea and vomiting (PONV) will be recorded. Vital signs will be measured for 15 minute intervals until criteria for discharge is met. A post-operative numeric pain score will be determined when the subject is ready for PACU discharge. On post operative day one, a follow up phone call will be made to the subject. He or she will be questioned as to their pain score and the use of pain medication since discharge.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing lower extremity surgery which requires the use of an inflated tourniquet ASA rating I-III

Exclusion Criteria:

* Allergy to alpha 2 adrenergic agonists
* Uncontrolled hypertension (SBP>180mm HG, Diastolic Blood Pressure >110mmHG)
* Heart block greater than first degree or cardiac muscle at risk for reversible ischemia
* Airway anatomy that contra-indicates the use of a laryngeal airway mask expected tourniquet time less than 60 minutes or greater than 150 minutes
* Subjects who do not have a phone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
hemodynamic stability | mean arterial pressure, heart rate and respiratory rate prior to surgery and at 5 minute intervals during surgery. same assessment in PACU until ready for discharge from PACU

SECONDARY OUTCOMES:
markers for stress response | prior to tourniquet inflation, 60 minutes after tourniquet inflation, 120 minutes after tourniquet inflation and 30 minutes after tourniquet release.

CONTACTS AND LOCATIONS:
Overall Officials: Jay S Berger, MD, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- New Jersey Medical School, Newark, New Jersey, United States